CLINICAL TRIAL: NCT06407739
Title: Effects of Three Phase Physical Therapy on Functional Activity in Children With Relapsed Club Foot After Ponseti Treatment
Brief Title: Three Phase Physical Therapy in Children With Relapsed Club Foot After Ponseti Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0770
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2025-03-12 (Actual); Status verified 2025-03

CONDITIONS: Club Foot
Keywords: Club foot; Ponseti technique; Three-phase physical therapy
MeSH Terms: conditions — Clubfoot

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Three-Phase Physical Therapy Intervention (Experimental): This group will be given the three-phase physical therapy intervention and each phase prolong for period of one month
  Interventions: Other: Three-Phase Physical Therapy Intervention

INTERVENTIONS:
Other: Three-Phase Physical Therapy Intervention — Phase 1: It include subtalar and talocrural joint mobilization in the supine position along with stretching and home education Stage 2: It include subtalar and talocrural joint mobilization in the supine position along with Kinesiotaping and functional exercises Phase 3: this phase include balance and propioceptive training aling with along with strengthening exercises of peroneal and tibialis anterior

SUMMARY:
Clubfoot, or congenital Talipes Equinovarus (CTEV), is a condition where a baby is born with one or both feet twisted inward and downward due to abnormal fetal foot development. Its estimated global prevalence is 1 in 1,000 live births, varying across populations. Relapsed clubfoot, a recurrence after initial correction, may occur due to incomplete treatment, noncompliance, muscle imbalance, or natural growth. Treatment involves surgical and non-surgical interventions, including soft tissue releases, osteotomies, and external fixation devices. The Ponseti method, a non-surgical approach, is commonly used in infants, with post-treatment physiotherapy focusing on three phases to optimize foot function. This holistic approach aims to achieve the best long-term outcomes for children with clubfoot. This 6-month randomized clinical trial at PSRD Hospital aims to assess the effectiveness of three-phase physical therapy versus conventional physiotherapy in treating clubfoot. With a sample size of 19 participants and a 10% attrition rate, the study involves children aged 3-10 previously treated with the Ponseti method. Data collection includes, one-leg standing and sit-to stand tests, Pirani score and the Oxford Ankle Foot Questionnaire. The three-phase therapy consists of joint mobilization, kinesio taping, and functional exercises over three months, with a focus on improving balance and proprioception.

ELIGIBILITY:
Inclusion Criteria:

* Having unilateral and bilateral club foot
* Age between 3-10 year
* Previously treated with Ponseti method
* Children fall under Grade II and III according to classification of relapse pattern

Exclusion Criteria:

* Children who were diagnosed with arthrogryposis multiplex congentia
* Children with spastic Equinovarus
* Children who had multiple surgical operation

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 19 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-08-05 (Actual); Study Completion 2024-09-15 (Actual)

PRIMARY OUTCOMES:
One leg standing test for Functional Activity | Baseline and 12th Week
  The one leg standing test is considered to be potentially useful for predicting functional deterioration. In the present study, we used the one leg standing test in the eyes open condition. The reliability of the SLS test is 0.89 and 0.86 with eyes opene
Sit to stand test for Functional Activity | Baseline and 12th Week
  The number of bilateral squats completed in 60 s is recorded

SECONDARY OUTCOMES:
Pirani score for Clubfoot Severity | Baseline and 12th Week
  PirS assesses six clinical signs characterizing clubfoot, three items for the midfoot, and three for the Hindfoot: medial crease (MC-Pir), lateral part of the head of the talus, the curvature of the lateral border, posterior crease, empty heel, and rigid equinus. Each of the six items are scored on a three-point scale (0 = none, 0.5 = moderate, 1 = severe abnormality). The total score ranges from 0 to 6 based on the severity of the deformity of the examined foot.
The oxford Ankle Foot questionnaire for children and parent for Functional Status | Baseline and 12th Week
  OxAFQ is a child or parent-reported (or caregiver) self-report health status questionnaire. (The Oxford Ankle Foot Questionnaire for Children (OxAFQ-C) - A Guide to the Scoring System, Oxford University Innovation Limited 2011). In this study, children and their parents were individually questioned

CONTACTS AND LOCATIONS:
Overall Officials: Fareeha Kausar, Principal Investigator — Riphah International University, Lahore, Pakistan
Locations (1):
- pakistan Society for the Rehabilitaion of Disables, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bent MA. Congenital Talipes Equinovarus (Clubfoot). Orthopaedics for the Newborn and Young Child: A Practical Clinical Guide: Springer; 2023. p. 47-60.
- [Background] Novotny T, Eckhardt A, Knitlova J, Doubkova M, Ostadal M, Uhlik J, Musilkova J. Increased Microvessel and Arteriole Density in the Contracted Side of the Relapsed Clubfoot. J Pediatr Orthop. 2020 Nov/Dec;40(10):592-596. doi: 10.1097/BPO.0000000000001563. PMID 32379245
- [Background] Grin L, van der Steen MC, Wijnands SDN, van Oorschot L, Besselaar AT, Vanwanseele B. Forefoot adduction and forefoot supination as kinematic indicators of relapse clubfoot. Gait Posture. 2021 Oct;90:415-421. doi: 10.1016/j.gaitpost.2021.09.185. Epub 2021 Sep 20. PMID 34583148
- [Background] Masrouha K, Chu A, Lehman W. Narrative review of the management of a relapsed clubfoot. Ann Transl Med. 2021 Jul;9(13):1102. doi: 10.21037/atm-20-7730. PMID 34423014